CLINICAL TRIAL: NCT00003185
Title: Adoptive Immunotherapy of Glioblastoma Multiforme With Tumor-Sensitized, Ex Vivo Activated T Lymphocytes
Brief Title: Biological Therapy in Treating Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066013; CCF-BB-IND-6154; NCI-H98-0008
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — FANG vaccine; sargramostim; Cyclophosphamide

INTERVENTIONS:
Biological: autologous tumor cell vaccine
Biological: sargramostim
Biological: tumor-draining lymph node lymphocyte therapy
Drug: cyclophosphamide
Procedure: conventional surgery

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase II trial to study the effectiveness of biological therapy in treating patients with glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the time to progression in patients with glioblastoma multiforme or anaplastic astrocytoma (primary presentation) treated with surgical resection, radiotherapy, and T cell immunotherapy as initial therapy. II. Determine the toxic effects of this therapy in these patients.

OUTLINE: Patients are vaccinated with irradiated, autologous tumor cells plus sargramostim (GM-CSF) intradermally near draining lymph nodes in the groin or axillary regions. This is then followed by 3 consecutive days of intradermal injections of GM-CSF only, directly into the vaccine sites. Enlarged lymph nodes are then removed 7-10 days later and activated with staphylococcal enterotoxin A (SEA) and interleukin-2 (IL-2). T cells are expanded ex vivo over approximately 10 days. 1-2 days prior to infusion, oral cyclophosphamide is administered as a one time dose. The lymphocyte infusion is then administered intravenously. Based on availability, patients may receive vaccine boosts with additional injections of irradiated autologous tumor cells thawed from the original, cryopreserved collection. Patients are followed at 1 month and then every 2 months thereafter.

PROJECTED ACCRUAL: A maximum of 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven glioblastoma multiforme or anaplastic astrocytoma Prior surgical resection and radiotherapy completed approximately 1 month prior to study

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-1 OR Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC greater than 2000/mm3 Platelet count greater than 100,000/mm3 Hepatic: No active infection with hepatitis B Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception during and for 1 month after study No active collagen vascular or autoimmune disease No prior severe reaction to any blood product No other prior malignancy within the past 5 years except adequately treated squamous cell or basal cell skin cancer, carcinoma in situ or the cervix, or stage I or II cancer in complete remission Not immunologically compromised due to chronic conditions Not allergic by standard skin testing HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy with immunomodulatory effects (e.g., interleukin-2, interferon alfa) Chemotherapy: No prior or concurrent local or systemic chemotherapy Endocrine therapy: At least 1 week since prior corticosteroid therapy No concurrent corticosteroid therapy Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Other: No concurrent antiproliferatives or immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1997-08; Study Completion 1998-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suyu Shu, PhD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Plautz GE, Barnett GH, Miller DW, Cohen BH, Prayson RA, Krauss JC, Luciano M, Kangisser DB, Shu S. Systemic T cell adoptive immunotherapy of malignant gliomas. J Neurosurg. 1998 Jul;89(1):42-51. doi: 10.3171/jns.1998.89.1.0042. PMID 9647171